CLINICAL TRIAL: NCT00077259
Title: A Phase II Study Of KOS-862 (Epothilone D), Administered Intravenously Weekly For 3 Weeks Every 4 Weeks, In The Second-Line Treatment Of Patients With Advanced Or Metastatic Colorectal Carcinoma (CRC)
Brief Title: Epothilone D as Second-Line Treatment for Patients With Advanced or Metastatic Refractory Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 03-113; MSKCC-03113; ROCHE-NO17320
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; recurrent rectal cancer; stage III colon cancer; stage III rectal cancer; stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — desoxyepothilone B

INTERVENTIONS:
Drug: epothilone D

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as epothilone D work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well epothilone D works as second-line therapy in treating patients with advanced or metastatic refractory colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of epothilone D as second-line treatment, in terms of objective response rate, in patients with advanced or metastatic refractory colorectal cancer.

Secondary

* Determine the safety of this drug in these patients.
* Determine the response duration in patients responding to treatment with this drug.
* Determine time to tumor progression and overall survival in patients treated with this drug.
* Correlate efficacy and safety with plasma concentrations of this drug and its major metabolites in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive epothilone D IV over 90 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 19-69 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced or metastatic adenocarcinoma of the colon or rectum
* Evidence of at least 1 site of unidimensionally measurable disease by radiography or physical examination
* Failed 1 prior treatment with a fluoropyrimidine in combination with either irinotecan OR oxaliplatin for advanced or metastatic disease
* No known CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin ≥ 9 g/dL
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (5 times ULN if hepatic metastases are present)
* Alkaline phosphatase ≤ 5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No New York Heart Association class III or IV congestive heart failure
* No QTc > 450 msec for males or > 470 msec for females
* No personal or family history of congenital long QT syndrome

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No pre-existing neuropathy grade 2 or greater
* No documented grade 3 or 4 hypersensitivity reaction to prior therapy containing Cremophor
* No infection requiring parenteral or oral anti-infective treatment
* No altered mental status or psychiatric condition that would preclude giving informed consent
* No other medical condition that would preclude study participation
* No other malignancy within the past 5 years except cured basal cell skin cancer, carcinoma in situ of the cervix or bladder, or stage T1 or T2 prostate cancer with a prostate-specific antigen < 2 ng/mL

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent sargramostim (GM-CSF)
* No concurrent routine prophylactic use of filgrastim (G-CSF)

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered

Endocrine therapy

* Not specified

Radiotherapy

* At least 3 weeks since prior radiotherapy and recovered

Surgery

* At least 3 weeks since prior surgery and recovered

Other

* More than 3 weeks since prior investigational agents (therapeutic or diagnostic)
* No other concurrent therapy for advanced or metastatic colorectal cancer
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10; Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B. Saltz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States